CLINICAL TRIAL: NCT00950625
Title: Comparison of Analgesic Efficacy of Intra-peritoneal Lignocaine With Bupivacaine After Laparoscopic Cholecystectomy: A Prospective Randomized Controlled Trial
Brief Title: Intraperitoneal Analgesia After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Muhammad Rizwan Khan, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 091026SUR
Record Dates: First submitted 2009-07-31; First posted 2009-08-03 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2009-07

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: intraperitoneal analgesia; laparoscopic cholecystectomy; lignocaine; bupevacaine
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- intraperitoneal lignocaine (Active Comparator): Intraperitoneal lignocaine will be compared with intraperitoneal bupevacaine for pain control after laparoscopic cholecystectomy
  Interventions: Drug: lignocaine; Drug: bupevacaine
- intraperitoneal bupevacaine (Active Comparator): intraperitoneal lignocaine will be compared with intraperitoneal bupevacaine after laparoscopic cholecystectomy
  Interventions: Drug: lignocaine; Drug: bupevacaine

INTERVENTIONS:
Drug: lignocaine — 200 mg of intraperitoneal lignocaine will be given once during surgery
Drug: bupevacaine — 100 mg of bupevacaine will be given once during laparoscopic cholecystectomy

SUMMARY:
Although laparoscopic cholecystectomy is associated with less pain than contemporary open procedures; it is definitely not pain free and the magnitude of postoperative shoulder and abdominal pain in the early postoperative period is still quite significant. This postoperative pain is a major concern not only for the patients, but also healthcare workers; and it often contributes to overnight hospital stay after this minimally invasive surgical procedure. Intraperitoneal instillation of local anesthetics at the time of surgery to control pain after laparoscopic cholecystectomy has been extensively studied in numerous randomized trials and found to be extremely useful. Lignocaine and Bupivacaine are two commonly used local anesthetic agents. In view of contradictory results from previous studies, it is not yet clear which of these two agents is superior to the other for pain control in this setting. To answer this question, we have designed a prospective randomized controlled trial and the specific aim of the study is to compare the analgesic efficacy of intraperitoneal lignocaine with intraperitoneal Bupivacaine in the postoperative setting after laparoscopic cholecystectomy.

If we can improve pain control after this minimally invasive procedure, it might result in decreased postoperative requirement of narcotic analgesia and its associated side-effects. It may also result in early recovery and the same day discharge of the patients with significant cost-containment for the patient and healthcare systems in future.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of symptomatic gallstones requiring laparoscopic cholecystectomy
* Elective surgical procedure
* American Society of Anesthesiologists class I and II

Exclusion Criteria:

* Patients refusing randomization
* Patients already on analgesics
* Patients with acute cholecystitis
* Patients requiring preoperative cholangiogram or common bile duct exploration
* Patients having bile or stone spillage during procedure
* Patients requiring conversion to open procedure
* Patients requiring re-exploration for any reason
* Patients with history of allergy to local anesthetic agents

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Pain Control after Laparoscopic Cholecystectomy | 24 hours after surgery

SECONDARY OUTCOMES:
Requirement of Analgesia after laparoscopic cholecystectomy | 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad R Khan, FRCS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan